CLINICAL TRIAL: NCT03077529
Title: Impact of Galacto-oligosaccharides on Microbial Fermentation Capacity and Markers of Frailty in Healthy Adults and Elderly
Brief Title: GOS and Microbial Fermentation in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 163046
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-04

CONDITIONS: Healthy Young Adults; Prefrail Elderly
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Galacto-oligosaccharide (Experimental): During this period subjects will receive 5.65 grams of Vivinal GOS supplements three times daily for four weeks
  Interventions: Dietary Supplement: Galacto-oligosacchride
- Maltodextrin (Placebo Comparator): During this period subjects will receive 7.24 grams of maltodextrin supplements three times daily for four weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Galacto-oligosacchride — During this period subjects will receive 5.65 grams of Vivinal GOS supplements three times daily for four weeks
  Arms: Galacto-oligosaccharide
Dietary Supplement: Maltodextrin — During this period subjects will receive 7.24 grams of maltodextrin supplements three times daily for four weeks
  Arms: Maltodextrin

SUMMARY:
The population is aging worldwide, concomitant frailty is increased in older age groups. Frailty has a strong impact on outcomes of multi-morbidity and daily living, thereby negatively influencing quality of life and health care costs. Prevention or delay of onset of frailty associated with aging is needed. Dietary intake of galacto-oligosaccharides (GOS) may have beneficial effects on microbiota composition and health outcome parameters. As microbiota composition and function may be altered in elderly compared to younger adults, it will investigated whether the effects of GOS on selected parameters of microbiota and gut health differ between elderly versus younger adults. The primary objective of this study is to compare the effects of four weeks GOS supplementation on intestinal microbiota composition and activity in elderly versus younger adults. Further, this study has four secondary objectives. The study conforms to a randomized double-blind placebo-controlled cross-over design per age-group. Study populations are human volunteers (male and female), healthy young adults of 25-50 years and prefail older adults of 70-85 years old, BMI 20-30 kg/m2. One intervention period subjects will receive 7.2 grams of Vivinal® GOS Powder three times daily for four weeks. The other intervention period subjects will receive isocaloric placebo supplements (5.7 grams maltodextrin) three times daily for four weeks. At the start and end of each intervention period, several measurements will take place. There will be a washout period of four to five weeks between intervention periods. The main study parameter is the change in microbial composition and activity induced by GOS intervention, in younger adults and elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Based on medical history no gastrointestinal complaints can be defined.
2. Age 25 - 50 years and classified as 'robust' by the Fried frailty criteria, or age 70 - 85 years and classified as 'prefrail' by the Fried frailty criteria.
3. Body Mass Index (BMI) ≥ 20 and < 30 kg/m2.
4. Weight-stable for at least 90 days prior to participation (no change in bodyweight, i.e. < 3kg).
5. Hemoglobin value of 8.2-11.0 mmol/L for men, 7.3-9.7 mmol/L for women.
6. C-reactive protein (CRP) value of <10 mg/L.
7. Creatinin value of 60-115 μmol/L for men, 50-100 μmol/L for women.
8. Alanine transaminase (ALAT) value of <45 U/L for men, 34 U/L for women.
9. Gamma-glutamyl transpeptidase (GGT) value of <55 U/L for men, <38 U/L for women.
10. Will be informed in case of any unexpected finding.

Exclusion Criteria:

1. History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol.
2. Self-admitted human immunodeficiency virus-positive state.
3. Disease with a life expectancy shorter than 5 years.
4. Abdominal surgery interfering with gastrointestinal function, upon judgment of the medical doctor, who will decide on in- or exclusion based on the surgery applied.
5. Use of antibiotics products within 90 days prior to the study.
6. Use of other medication will be reviewed by a medical doctor, who will decide on in- or exclusion based on the drug(s) used.
7. Use of laxatives within 14 days prior to the study.
8. Institutionalized (e.g. hospital or nursing home).
9. Pregnancy or lactation.
10. Plan to lose weight or follow a specific diet within the study period.
11. Alcohol intake >14 units/week.
12. Drug use.
13. Blood donation within 30 days prior to the study.
14. Administration of probiotic or prebiotic supplements, investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principle investigator), in the 14 days prior to the study.
15. History of side effects towards intake of prebiotic supplements.
16. Self-admitted lactose intolerance

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Microbial composition | Change from baseline to four weeks supplementation, of each intervention period
  Microbiota composition and functional capacity as measured by HiSeq sequencing of fecal 16S rRNA genes.
Microbial activity | Change from baseline to four weeks supplementation, of each intervention period
  Microbial activity as measured by metabolites, such as organic acids analysis in feces and plasma.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilms E, An R, Smolinska A, Stevens Y, Weseler AR, Elizalde M, Drittij MJ, Ioannou A, van Schooten FJ, Smidt H, Masclee AAM, Zoetendal EG, Jonkers DMAE. Galacto-oligosaccharides supplementation in prefrail older and healthy adults increased faecal bifidobacteria, but did not impact immune function and oxidative stress. Clin Nutr. 2021 May;40(5):3019-3031. doi: 10.1016/j.clnu.2020.12.034. Epub 2021 Jan 12. PMID 33509667